CLINICAL TRIAL: NCT01542788
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of GS-7977 + Ribavirin for 12 Weeks in Subjects With Chronic Genotype 2 or 3 HCV Infection Who Are Interferon Intolerant, Interferon Ineligible or Unwilling to Take Interferon
Brief Title: Sofosbuvir + Ribavirin for 12 Weeks in Subjects With Chronic Genotype 2 or 3 Hepatitis C Infection Who Are Interferon Intolerant, Interferon Ineligible or Unwilling to Take Interferon
Acronym: POSITRON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-334-0107
Record Dates: First submitted 2012-02-17; First posted 2012-03-02 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Hepatitis C
Keywords: HCV genotype 2 (GT-2); HCV genotype 3 (GT-3); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Interferon intolerant; Interferon ineligible; GS-7977; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF+RBV (Experimental): Participants were randomized to receive SOF+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Placebo (Placebo Comparator): Participants were randomized to receive placebo to match SOF plus placebo to match RBV for 12 weeks.
  Interventions: Drug: Placebo to match SOF; Drug: Placebo to match RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: SOF+RBV
Drug: RBV — Ribavirin (RBV) was administered as a tablet orally according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg).
  Arms: SOF+RBV
Drug: Placebo to match SOF — Placebo to match SOF was administered orally once daily.
  Arms: Placebo
Drug: Placebo to match RBV — Placebo to match RBV was administered orally twice daily.
  Arms: Placebo

SUMMARY:
This multicenter study was to evaluate subjects with chronic genotype 2 or 3 HCV infection who were interferon (IFN) ineligible, IFN intolerant or unwilling to take IFN. Participants were randomized in a 3:1 ratio to receive sofosbuvir (SOF)+ribavirin (RBV), or placebo to match SOF+placebo to match RBV. Randomization was stratified by presence/absence of cirrhosis. Approximately 20% of participants may have had evidence of cirrhosis at screening.

DETAILED DESCRIPTION:
Participants who were randomized to the placebo arm and completed all scheduled study procedures were eligible to receive active SOF+RBV in open-label Study GS-US-334-0109.

Participants who do not achieve sustained virologic response (SVR) were eligible for enrollment in the Sequence Registry Study GS-US-248-0123. The purpose of the Sequence Registry Study is to monitor the persistence of resistant mutations for up to 3 years.

Participants who achieved SVR were eligible for enrollment in the SVR Registry Study GS-US-248-0122. The purpose of the SVR Registry Study is to evaluate durability of SVR for up to 3 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infection with HCV genotype 2 or 3
* Cirrhosis determination
* Subject meets one of the following classifications:

  1. IFN unwilling
  2. IFN ineligible
  3. IFN intolerant
* Screening laboratory values within defined thresholds
* Subject has not been treated with any investigational drug or device within 30 days of the Screening visit
* Use of highly effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Prior exposure to an direct-acting antiviral targeting the HCV nonstructural protein (NS)5B polymerase
* Pregnant or nursing female or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Excessive alcohol ingestion or significant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (50):
  - University of Alabama Birmingham, Birmingham, Alabama
  - SCTI Research Foundation Liver Center, Coronado, California
  - Kaiser Permanente, Los Angeles, California
  - Lightspeed Medical, Los Angeles, California
  - Anthony Mills MD, Inc., Los Angeles, California
  - Medical Associates Research Group, San Diego, California
  - UCSD Antiviral Research Center, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami, Center for Liver Diseases, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Orlando Immunology Center (ACH), Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - ID Care, Hillsborough, New Jersey
  - Binghamton Gastroenterology Associates, Binghamton, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Inova Fairfax Hospital Center for Liver Diseases, Falls Church, Virginia
  - Liver Institute of Virginia, Bon Secours St.Mary's, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - St. Vincent's Hospital, Melbourne
  - Monash Medical Centre, Melbourne
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - (G.I.R.I.) Gastrointestinal Research Institute, Vancouver, British Columbia
  - Toronto Liver Centre, Toronto, Ontario
  - CHUM - The Research Centre, Montreal, Quebec
- New Zealand (2):
  - Auckland Clinical Studies Limited, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - Fundacion De Investigacion De Diego, San Juan, Puerto Rico
  - Clinical Research Puerto Rico Inc, San Juan

REFERENCES:
- [Derived] Stepanova M, Nader F, Cure S, Bourhis F, Hunt S, Younossi ZM. Patients' preferences and health utility assessment with SF-6D and EQ-5D in patients with chronic hepatitis C treated with sofosbuvir regimens. Aliment Pharmacol Ther. 2014 Sep;40(6):676-85. doi: 10.1111/apt.12880. Epub 2014 Jul 15. PMID 25040192
- [Derived] Jacobson IM, Gordon SC, Kowdley KV, Yoshida EM, Rodriguez-Torres M, Sulkowski MS, Shiffman ML, Lawitz E, Everson G, Bennett M, Schiff E, Al-Assi MT, Subramanian GM, An D, Lin M, McNally J, Brainard D, Symonds WT, McHutchison JG, Patel K, Feld J, Pianko S, Nelson DR; POSITRON Study; FUSION Study. Sofosbuvir for hepatitis C genotype 2 or 3 in patients without treatment options. N Engl J Med. 2013 May 16;368(20):1867-77. doi: 10.1056/NEJMoa1214854. Epub 2013 Apr 23. PMID 23607593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 54 sites in the North America, Australia, and New Zealand. The first participant was screened on 07 March 2012. The last participant observation was on 04 February 2013.
Pre-assignment Details: 410 participants were screened and 280 were randomized. Of those participants randomized, 278 received at least one dose of study drug, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- SOF+RBV: Participants were randomized to receive sofosbuvir (SOF)+ribavirin (RBV) for 12 weeks. SOF was administered as a 400 mg tablet orally once daily. RBV was administered as 200 mg tablets (1000-1200 mg daily based on weight) according to package insert recommendations.
- Placebo: Participants were randomized to receive placebo to match SOF plus placebo to match RBV for 12 weeks. Placebos were administered in the same manner as their active counterparts.
Period: Overall Study
Arm/Group | SOF+RBV | Placebo
Started | 209 | 71
Randomized and Treated | 207 | 71
Completed | 154 | 0
Not Completed | 55 | 71
Not completed — Randomized but Not Treated | 2 | 0
Not completed — Lack of Efficacy | 41 | 71
Not completed — Lost to Follow-up | 5 | 0
Not completed — Death | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the Safety Analysis Set (randomized and received at least 1 dose of study drug) were analyzed for baseline characteristics.
Groups:
- SOF+RBV: Participants were randomized to receive SOF+RBV for 12 weeks. SOF was administered as a 400 mg tablet orally once daily. RBV was administered as 200 mg tablets (1000-1200 mg daily based on weight) according to package insert recommendations.
- Total: Total of all reporting groups
Arm/Group | SOF+RBV | Placebo | Total
Number analyzed (Participants) | 207 | 71 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9.9) | 52 (8.2) | 52 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 37 | 127
  Male | 117 | 34 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 11 | 30
  Not Hispanic or Latino | 188 | 60 | 248
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 4 | 13
  White | 188 | 66 | 254
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 168 | 60 | 228
  Canada | 15 | 8 | 23
  Australia | 18 | 3 | 21
  New Zealand | 6 | 0 | 6
Cirrhosis [Number; unit: participants]
  No | 176 | 58 | 234
  Yes | 31 | 13 | 44
HCV Genotype [Number; unit: participants]
  Genotype 2 | 109 | 34 | 143
  Genotype 3 | 98 | 37 | 135
IL28 Genotype [Number; unit: participants]
  CC | 97 | 29 | 126
  CT | 84 | 36 | 120
  TT | 26 | 6 | 32
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.77) | 6.3 (0.76) | 6.3 (0.77)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 67 | 17 | 84
  ≥ 6 log10 IU/mL | 140 | 54 | 194
Interferon Classification [Number; unit: participants]
  Ineligible | 88 | 33 | 121
  Intolerant | 17 | 8 | 25
  Unwilling | 102 | 30 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving SVR12
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ, ie, < 25 IU/mL) 12 weeks after cessation of therapy
Time Frame: Post-treatment Week 12
Population: Full Analysis Set: participants with genotype 2 or 3 HCV infection who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | Placebo
Number analyzed (Participants) | 207 | 71
percentage of participants | 78 | 0
Statistical Analysis 1: Comparison: SOF+RBV vs Placebo; A sample size of 180 subjects in the active group and 60 in the placebo group would provide 99% power to detect a difference between group SVR12 rates of 40% using a 2-sided continuity-corrected chi-square test at significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is from the Cochran-Mantel-Haenszel test stratified by presence or absence of cirrhosis for the superiority of SOF+RBV over placebo; Proportion difference = 77.3, 95% CI 2-sided [71.0 to 83.6] — The difference in proportions between treatment groups and associated 95% confidence interval (CI) are calculated based on stratum-adjusted Mantel-Haenszel proportions

2. Primary Outcome: Number of Participants Experiencing Adverse Events Leading to Permanent Discontinuation of Study Drug
Description: The number of subjects experiencing adverse events leading to permanent discontinuation of study drug was summarized. Adverse events may or may not have been related to study treatment.
Time Frame: Baseline to Week 12
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | SOF+RBV | Placebo
Number analyzed (Participants) | 207 | 71
participants
  No adverse event leading to discontinuation | 202 | 68
  Abdominal pain upper | 1 | 0
  Alanine aminotransferase increased | 0 | 1
  Anaemia | 1 | 0
  Anxiety | 1 | 0
  Chest discomfort | 1 | 0
  Injury | 1 | 0
  Insomnia | 1 | 0
  Muscle spasms | 1 | 0
  Oedema peripheral | 0 | 1
  Pancreatitis | 0 | 1
  Rash | 0 | 1
  Road traffic accident | 1 | 0

3. Secondary Outcome: Percentage of Participants Achieving SVR4
Description: SVR4 was defined as HCV RNA < LLOQ 4 weeks after cessation of therapy
Time Frame: Post-treatment Week 4
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | Placebo
Number analyzed (Participants) | 207 | 71
percentage of participants | 83.1 | 0.0
Statistical Analysis 1: Comparison: SOF+RBV vs Placebo; Test type: Superiority or Other; Proportion difference = 82.7, 95% CI 2-sided [76.8 to 88.5] — The difference in proportions between treatment groups and associated 95% CI are calculated based on stratum-adjusted Mantel-Haenszel proportions

4. Secondary Outcome: Percentage of Participants Achieving SVR24
Description: SVR24 was defined as HCV RNA < LLOQ 24 weeks after cessation of therapy
Time Frame: Post-treatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | Placebo
Number analyzed (Participants) | 207 | 71
percentage of participants | 77.8 | 0.0
Statistical Analysis 1: Comparison: SOF+RBV vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is from the Cochran-Mantel-Haenszel test stratified by randomization stratification factor for the superiority of SOF+RBV over placebo; Proportion difference = 77.3, 95% CI 2-sided [71.0 to 83.6] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants Experiencing Viral Breakthrough
Description: Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment, confirmed with 2 consecutive values (second confirmation value could be posttreatment), or last available on-treatment measurement with no subsequent follow-up values
Time Frame: Baseline to Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | Placebo
Number analyzed (Participants) | 207 | 71
percentage of participants | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: End of treatment to post-treatment Week 24
Population: Participants in the Full Analysis Set who had an end-of-treatment response (HCV RNA < LLOQ as the last observed on-treatment value) were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | Placebo
Number analyzed (Participants) | 205 | 0
percentage of participants | 20.5 |

ADVERSE EVENTS:
Time Frame: Baseline to last dose date of study regimen + 30 days
Arm/Group | SOF+RBV | Placebo
Serious Adverse Events (participants affected / at risk) | 11/207 | 2/71
Other Adverse Events (participants affected / at risk) | 184/207 | 55/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=207) | Placebo (N=71)
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=207) | Placebo (N=71)
Anaemia (Blood and lymphatic system disorders) | 27 | 0
Nausea (Gastrointestinal disorders) | 46 | 13
Diarrhoea (Gastrointestinal disorders) | 19 | 4
Vomiting (Gastrointestinal disorders) | 12 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Fatigue (General disorders) | 91 | 17
Irritability (General disorders) | 19 | 1
Oedema peripheral (General disorders) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 1
Headache (Nervous system disorders) | 43 | 14
Dizziness (Nervous system disorders) | 19 | 5
Insomnia (Psychiatric disorders) | 39 | 3
Anxiety (Psychiatric disorders) | 13 | 4
Depression (Psychiatric disorders) | 15 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 6
Rash (Skin and subcutaneous tissue disorders) | 18 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years